CLINICAL TRIAL: NCT01924988
Title: Prostate Embolization for Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: James B. Spies, MD (Other)
Responsible Party: Sponsor-Investigator, James B. Spies, MD, Chair, Department of Radiology, Georgetown University
Organization: Georgetown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G120110
Record Dates: First submitted 2013-08-14; First posted 2013-08-19 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH, benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostatic Embolization (Experimental): Therapeutic occlusion of the prostate arteries
  Interventions: Device: Prostatic Embolization with Embosphere Micropsheres

INTERVENTIONS:
Device: Prostatic Embolization with Embosphere Micropsheres — Each patient will have a selective internal iliac arteriogram, and as necessary, an arteriogram of the anterior division of the internal iliac artery performed to identify the prostatic arterial supply. This typically arises from the inferior vesicle artery (also known as the prostatic artery), but may have supply from the superior vesicle, the internal pudendal or obturator branches as well.
  The prostatic arteries will be selected using standard micro-catheter technique. Embolization of the prostate will be performed with 300 to 500 um sized TAGM (Embosphere® Microspheres, Merit Medical, South Jordan, UT). The embolization endpoint will be absence of the normal blush of the prostate on post embolization angiography and stasis of flow in the prostate arteries.

SUMMARY:
This is a Phase I/II investigator sponsored FDA-approved Investigational Device Exemption protocol, with the primary goal of determining the safety of prostatic artery embolization (PAE) for benign prostatic hyperplasia. Our primary goal is to document the frequency of side effects, particularly bladder and rectal complications, which may occur as a result of this procedure. Secondarily, the study will provide preliminary data to determine its effectiveness in diminishing obstructive symptoms associated with BPH.

DETAILED DESCRIPTION:
Objectives of the investigation

This study has a primary goal of determining the safety of prostatic artery embolization (PAE) for benign prostatic hyperplasia. Our primary outcome is the frequency of adverse events, particularly bladder and rectal complications, which may occur as a result of this procedure. Secondarily, the study will allow us to begin to determine its effectiveness in diminishing obstructive symptoms associated with BPH.

Duration of investigation

The investigation will enroll 30 patients, with a target enrollment period of less than 12 months. Each patient will be consented for follow-up up to 5 years, but each patient will reach the first important safety endpoint 1 week after treatment and the first clinical efficacy assessment 3 months after treatment.

Objectives

To determine the safety and effectiveness of prostate artery embolization for the treatment of BPH.

Description of study type

This is a prospective non-comparative treatment study of an initial cohort of 30 patients.

Study Population

The patients will be recruited from the urology practice at Georgetown University and from other urologists in the area and by patient self-referral. The study also will be announced on a study website, the content of which will be approved by the IRB at Georgetown University Medical Center.

The primary outcome is the absence of complications to the bladder, rectum or other pelvic structures detected in the first week after therapy. Each patient will be judged free of these adverse events or not. For those with an adverse event, the complication will be scored using the Society of Interventional Radiology (SIR) definitions. Descriptive statistics will be used to summarize these events, along with patient demographics and initial clinical status.

Appropriate parametric and non-parametric tests will be used to assess change in laboratory measures, urine flowmetry parameters, and scores from the IPSS and IIEF. Changes in prostate volumes and the estimated volume of devascularized tissue will be calculated for each patient and outcomes from the different embolics will be compared. Appropriate paired parametric and non-parametric tests will be used to determine statistical significance. A p value of 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. You must have symptoms from BPH for at least 6 months
2. Your symptoms must meet the entrance criteria, as determined by a short questionnaire you will be asked to complete.
3. You must have urinary flow rates that meet entrance criteria, as measured by a simple urination test.
4. Enlargement of the prostate, as measured by the urologist, with a volume of between 50 and 100 cc.
5. You must be at least 50 years of age, but not more than 90.

Exclusion Criteria:

* 1. Prostate Cancer 2. Blockage of major arteries in your pelvis or other arterial abnormalities that prevent embolization or that might increase risks of injury. You will be screened for these conditions if you consent to participate.

  3. Significantly decreased kidney function 4. Prior prostate surgery, whether it has been performed via a scope through the penis or with conventional surgery.

  5. Bladder or urinary conditions other than BPH requiring therapy. You will be screened for these conditions if you consent to participate.

  6. History of cardiac rhythm abnormalities, congestive heart failure, uncontrolled diabetes, significant respiratory disease, or known immunosuppression.

  7. History of clotting disorders. 8. Current medications (use of alpha-blockers within two months, 5-alpha-reductase inhibitors within six months, anti-cholinergics within two months, and beta blockers, antihistamines, anticonvulsants, or antispasmodics within one week of treatment unless you have been on the same drug with a stable urination pattern.

  9. Active urinary tract infection 10. Allergy to iodinated contrast agents, collagen or gelatin products 11. Acute urinary retention that has NOT been treated by a urinary catheter. 12. Significant retained urine after voiding as measured by ultrasound. In this case, significant means more than 250 ml (about 1 cup).

  13. Bladder stones or blood in urine within three months 14. Previous rectal surgery, excluding hemorrhoidectomy (removal of hemorrhoid), or history of rectal disease 15. Prior pelvic irradiation or radical pelvic surgery 16. If you are interested in future fertility 17. Unable to speak and read English.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostatic Embolization: This single-center, Phase I prospective, observational, non-comparative study of the safety and effectiveness of prostate artery embolization for symptomatic benign prostatic hyperplasia. The primary outcome was to determine the frequency of adverse events, focusing on procedure-related bladder and rectal complications as detected by cystoscopic and anoscopic assessment post-treatment. The secondary objectives were to measure the effectiveness in diminishing symptoms of lower urinary tract symptom (LUTS) from treatment.
  The inclusion criteria were as follows: Men presenting with benign prostatic hyperplasia with symptoms for at least 6 months. Additional criteria included moderate to severe obstructive urinary tract symptoms as defined as an International Prostate Symptom Score (IPSS) score of 12 or greater, and peak urinary flow (QMax) of less than 12 mL/s or acute urinary retention.
Period: Overall Study
Arm/Group | Prostatic Embolization
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety of Prostate Artery Embolization: This is a study focused on the safety of prostate artery embolization based primarily on cystoscopic evaluation after embolization.
Arm/Group | Safety of Prostate Artery Embolization
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 69.6 [59 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 15
Prostate Size [Mean (Full Range); unit: Grams] | 71.9 [51 to 99]
International Prostate Symptom Score (IPSS) score [Mean (Full Range); unit: units on a scale] — Validated patient reported questionnaire to assess the severity of lower urinary tract symptoms associated with benign prostatic enlargement. Scores range from 0 to 35, with a score of 0-7 considered mild, 8-19 moderate and 20 to 35 severe symptoms.
  units on a scale | 23.2 [12 to 35]
International index of erectile function- 5 (IIEF-5) score [Mean (Full Range); unit: units on a scale] — International index of erectile function- 5 is a sexual health of men (SHIM) validated 5 question questionnaire assessing erectile function and sexual function, with a range of scores from 5 to 25, higher scores indicating better erectile function.
  units on a scale | 12.2 [5 to 25]
Baseline Cystoscopy findings [Count of Participants; unit: Participants] — Those with normal cystoscopic findings prior to intervention
  Participants | 15
Maximum urinary flow [Mean (Full Range); unit: ml/sec] | 7.3 [2.6 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bladder or Rectal Injury
Description: Bladder injury as detected by cystoscopy. Rectal injury detected by anoscopy.
Time Frame: Evaluated 1 week after procedure
Population: 1 patient failed to complete this follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Prostate Artery Embolization: Therapeutic embolization of the prostate arteries to treat benign prostatic hyperplasia.
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 14
Participants | 0

2. Primary Outcome: Detection of Bladder Injury
Description: Bladder injury as detected by cystoscopy
Time Frame: 3 months after treatment
Population: 9 participants failed to complete this follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Prostate Artery Embolization: Therapeutic embolization of the prostate for treatment of benign prostate hyperplasia
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Detection of a Bladder Injury
Description: Bladder injury detected by cystoscopy
Time Frame: 6 months after treatment
Measure: Count of Participants; unit: Participants
Groups:
- Number With Bladder Injury at 3 Months: Those with bladder injury detected by cystoscopy
Arm/Group | Number With Bladder Injury at 3 Months
Number analyzed (Participants) | 7
Participants
  Patients evaluated | 7
  Number with bladder injury | 0

4. Primary Outcome: Detection of a Bladder Injury by Cystoscopy
Description: Number of patients with a bladder injury detected by cystoscopic examination
Time Frame: 12 months after the procedure
Measure: Count of Participants; unit: Participants
Groups:
- Cystoscopy Outcomes 12 Months: Number of patients with a bladder injury 12 months after treatment.
Arm/Group | Cystoscopy Outcomes 12 Months
Number analyzed (Participants) | 2
Participants
  Number evaluated | 2
  Number with bladder injury | 0

5. Secondary Outcome: International Prostate Symptom Score (IPSS)
Description: Measure Description: Validated patient reported questionnaire to assess the severity of lower urinary tract symptoms associated with benign prostatic enlargement. Severity of symptom scores range from 0 to 35, with a score of 0-7 considered mild, 8-19 moderate and 20 to 35 severe symptoms.
Time Frame: 1week, 3 months, 6months, 12months
Population: Some participants did not complete follow-up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 14
score on a scale
  1 week | 15.2 [3 to 29]
  3 months: number analyzed (Participants) | 10
  3 months | 9.1 [2 to 21]
  6 months | 9.5 [3 to 22]
  12 months: number analyzed (Participants) | 2
  12 months | 17.5 [17 to 18]

6. Secondary Outcome: International Index of Erectile Function (IIEF)- 5
Description: Measure Description: IIEF-5 is a 5 question validated patient reported outcome measure or erectile dysfunction (ED), with a range of scores from 5 to 25, and ED was classified into five categories or erectile function based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
Time Frame: 1week, 3 months, 6months, 12months
Population: Some participants did not complete follow-up
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 15
score on a scale
  1 week: number analyzed (Participants) | 7
  1 week | 17.3 [9 to 25]
  3 months: number analyzed (Participants) | 10
  3 months | 12.4 [5 to 24]
  6 months: number analyzed (Participants) | 8
  6 months | 11.9 [5 to 23]
  12 months: number analyzed (Participants) | 2
  12 months | 8 [7 to 9]

7. Secondary Outcome: QMax (Peak Urinary Flow)
Description: Measure Description: measure of the peak urinary flow rate as measured by urine flowmetry. Result is in ml/sec.
Time Frame: 1week, 3 months, 6months, 12months
Population: Some participants did not complete follow-up
Measure: Mean (Full Range); unit: milliliters per second
Arm/Group | Prostate Artery Embolization
Number analyzed (Participants) | 15
milliliters per second
  1 week: number analyzed (Participants) | 7
  1 week | 10.4 [0 to 21]
  3 months: number analyzed (Participants) | 3
  3 months | 18.1 [6.8 to 37.8]
  6 months: number analyzed (Participants) | 4
  6 months | 10.4 [2 to 12.1]
  12 months: number analyzed (Participants) | 1
  12 months | 2.2 [2.2 to 2.2]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Society of Interventional Radiology Adverse Events Classification Class A Minor, no treatment Class B Minor, medical or nominal therapy Class C Major, re-admission for less than 48 hrs, ED visit, minor intervention Class D Major, re-admission for greater than 48 hrs, major intervention Class E Major, permanent patient injury Class F Major, patient death
Groups:
- Adverse Events: Summary of adverse events
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 10/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=15)
Dysuria or urethral pain (Renal and urinary disorders) | 6 (6)
Hematuria (Renal and urinary disorders) | 1 (1) — Self limited blood in urine
acute prostatitis (Renal and urinary disorders) | 1 (1) — Prostate tenderness, dysuria, and positive urinary culture
Reported fever and chills (Renal and urinary disorders) | 1 (1) — Fever and chills reported but without infection, not documented by research staff
Headache and confusion (Nervous system disorders) | 1 (1) — Headache and confusion reported but not documented by research staff

LIMITATIONS AND CAVEATS:
There as poor compliance by patients to the follow-up protocol beyond 1 week post procedure. Only 10 of 15 patients participated in follow-up at three months. By 12 months, only 3 patients provided some elements of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT01924988/Prot_SAP_000.pdf